CLINICAL TRIAL: NCT07166016
Title: Evaluating the Effectiveness of Treatments on Gait Biomechanics in Patients With Hammertoe Deformities
Brief Title: Treatment Effects on Gait in Hammertoe Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Rio Grande Valley (Other)
Responsible Party: Principal Investigator, Hafizur Rahman, Assistant Professor, University of Texas Rio Grande Valley
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-24-0101
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Hammertoe
Keywords: Hammertoe; Plantar pressure
MeSH Terms: conditions — Hammer Toe Syndrome | interventions — Conservative Treatment; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conservative Treatment (Experimental)
  Interventions: Other: Conservative
- Surgical Treatment (Experimental)
  Interventions: Procedure: Surgical

INTERVENTIONS:
Other: Conservative — Patients with hammertoe deformities will undergo conservative treatments, including wearing proper shoes, insoles, and custom orthotics.
  Arms: Conservative Treatment
Procedure: Surgical — Patients with hammertoe deformities will undergo surgical treatments.
  Arms: Surgical Treatment

SUMMARY:
This study looks at how hammertoe deformities affect foot pressure distribution and whether proper treatment can improve quality of life.

DETAILED DESCRIPTION:
Hammertoe deformities often lead to pain, discomfort, and difficulty with walking. People affected by these deformities are also at a higher risk for developing pressure-related ulcers on their feet. It is essential for clinicians to be aware of this risk and to assess the degree of plantar pressure reduction following both conservative and surgical treatments, as alleviating this pressure may help prevent the development of foot ulcers. Individuals diagnosed with hammertoes will participate in two data collection sessions-one visit before the intervention begins (pre-intervention) and another visit three months after the intervention (post-intervention).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed distal symmetric sensory neuropathy.
* MTPJ hyperextension deformity.
* Claw or hammer toe deformity in toes.

Exclusion Criteria:

* Non-hammertoe foot deformities affecting metatarsal head pressure.
* Limited joint mobility, lower-limb amputation, or Charcot neuro-osteoarthropathy.
* Peripheral vascular disease
* Non-diabetic neuropathies
* Significant lower-limb musculoskeletal issues
* Rheumatoid arthritis
* Current foot ulcer or edema
* Inability to walk unaided
* MRI contraindications
* Morton's neuroma
* History of foot surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
In-shoe Peak Plantar Pressure | Pre-intervention, Post-intervention (3 months)
  In-shoe peak plantar pressure data will be recorded as patients walk with a pressure-measuring sensor placed inside their shoes. The unit will be Kilopascal (kPa).

SECONDARY OUTCOMES:
Quality of Life Questionnaire | Pre-intervention, Post-intervention (3 months)
  Medical Outcomes Study 36-item Short Form questionnaires (SF-36) will be used to assess the quality of life. The SF-36 form has four subsections: pain, distance, walking speed, and stair climbing. Each subsection score ranges from 0 to 100 (where 0 is the worst, and 100 is the best health status).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Rio Grande Valley, Harlingen, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified and anonymous dataset will be created for sharing purposes. The dataset will only be shared upon reasonable request and with a written agreement from the recipient. All outcomes, results, and findings will be published in peer-reviewed journals and conference proceedings.
Time Frame: The de-identified and anonymous dataset will only be shared after the study is completed and results are published in peer-reviewed journals and conference proceedings.